CLINICAL TRIAL: NCT02071095
Title: Simultaneous Disruption of Latency and Immune Enhancement by Poly-ICLC During HIV-1 Infection
Brief Title: Enhancement by Poly-ICLC During HIV-1 Infection
Acronym: Poly-ICLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nina Bhardwaj (Other)
Collaborators: The Campbell Foundation (Other); Oncovir, Inc. (Industry); National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Nina Bhardwaj, Professor, Medicine - Director, Immunotherapy Program, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 13-0482; Campbell Foundation (Other Grant/Funding Number: Campbell Foundation); 1R21AI110736-01 (NIH)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: HIV-1 Infected Adults With Chronic HIV-1 Infection
Keywords: Human immunodeficiency virus 1; Combined Antiretroviral Therapy; Poly-ICLC; Adjuvant
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — poly ICLC

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Poly-ICLC (Experimental): Arm A (N=15): Patients will receive an injection of 1.4 mg of Poly-ICLC (Hiltonol®, Oncovir) subcutaneously on day 1 and day 2.
  Interventions: Drug: Arm A: Poly-ICLC
- Arm B: Normal Saline (Placebo Comparator): Arm B: (N=5): Patients will receive an injection of normal saline subcutaneously on day 1 and day 2.
  Interventions: Drug: Arm B: Normal Saline

INTERVENTIONS:
Drug: Arm A: Poly-ICLC — Poly-ICLC (Hiltonol®, Oncovir) Administration - On days 1 and 2, patients randomized to this arm will be injected subcutaneously in the arm with 1.4 mg of Poly-ICLC (Hiltonol®, Oncovir). Each subject will receive a total of 2 SC doses of Poly-ICLC. The volume of each injection is 0.7ml. The investigators who are blinded will not be present at the time of injection by the study nurse.
  Other Names: Poly-ICLC (Hiltonol®, Oncovir)
  Arms: Arm A: Poly-ICLC
Drug: Arm B: Normal Saline — Normal Saline - On days 1 and 2, patients randomized to this arm will be injected subcutaneously in the arm with normal saline obtained from the Rockefeller University Pharmacy. Each subject will receive a total of 2 SC doses of normal saline. The volume of each injection is 0.7ml. The investigators who are blinded will not be present at the time of injection by the study nurse.
  Other Names: Placebo
  Arms: Arm B: Normal Saline

SUMMARY:
This study involves researching new approaches to treating HIV infection. Currently, HIV infection is treated with combinations of drugs called antiretrovirals. These drugs protect cells from infection by interfering with the viruses' ability to make copies of itself by infecting new target cells. Though these drugs are very effective, they cannot cure HIV infection and must be taken each and every day at prescribed doses to maintain their beneficial effect. This research study is investigating a new approach that involves an addition to existing medications.

The study is investigating a medication called Poly-ICLC (Hiltonol®, Oncovir), which is an adjuvant. Adjuvants are medications that are designed to boost your body's immune responses resulting from a vaccine. The investigators want to test whether Poly-ICLC is an adjuvant that is effective in HIV-infected patients. A vaccine is not given in this study, but just investigating the adjuvant, Poly-ICLC, to determine whether it may be safe and useful in future vaccines that could be used to treat HIV, called therapeutic vaccines. One goal of future therapeutic vaccines is to reduce the virus that remains persistently inside of cells in a dormant or resting state despite treatment with HIV medications. This persistent pool is termed the "latent virus pool" or "viral reservoir". One tactic to reduce this viral reservoir is to first stimulate HIV to start replicating in order to force it out of hiding. Once viral replication occurs, the infected cells may then be recognized and killed by cells of the immune system. Therefore, we also want to see what effect Poly-ICLC has on the virus that lives inside of cells. Specifically, the investigators want to look at whether Poly-ICLC increases the level of virus inside your cells while also improving your immune system's responses.

The investigators are doing this research in hope to find new ways to treat HIV infection that may reduce exposure to medications that are called antiretrovirals. Antiretrovirals are medications used to treat HIV infection. They are very effective but have side effects and have to be taken each and every day and cannot cure HIV.

DETAILED DESCRIPTION:
Effective combination antiretroviral therapy (cART) has dramatically altered the morbidity and mortality associated with human immunodeficiency virus (HIV-1) infection. Nevertheless, the current treatment paradigm of lifelong antiviral therapy with near perfect patient adherence to avoid the emergence of drug resistant HIV remains less than ideal and this therapeutic approach has clear limitations.

In addition to long term toxicities associated with currently preferred therapies, combination therapy for HIV-1 infection cannot address the issue of viral persistence. HIV-1 persists in both blood and tissue despite long-term suppression with antiretroviral agents (ARVs). Eradication strategies for HIV-1 are likely to require a multi-faceted approach to reduce the latent reservoir, with key components focusing upon both the disruption of viral latency and the enhancement of cytotoxic T lymphocyte (CTL) function to promote killing of infected cells. In order to successfully achieve these objectives, agents that safely stimulate replication of the latent reservoir AND explore approaches to enhance HIV-specific adaptive immunity to augment CTL function must be investigated. The investigators propose that this may be accomplished with a single therapeutic modality that is devised appropriately. Certain adjuvants may possess immunostimulatory properties that trigger transient activation of viral transcription while simultaneously enhancing HIV-specific CTL function and, thus, may play an important role in such a vaccine.

Here, the investigators propose a proof of concept clinical trial to determine the ability of Poly-ICLC (Hiltonol®, Oncovir), to safely activate the latent viral reservoir and enhance innate immunity when administered to HIV-infected individuals. This randomized, double-blinded, placebo-controlled study will administer two doses of Poly-ICLC to HIV-infected individuals whom are virologically suppressed on combination anti-retroviral therapy (cART). The investigators hypothesize that Poly-ICLC will be safe and well-tolerated and will transiently disrupt viral latency while enhancing innate immune responses. Should this be the case, then Poly-ICLC would be an ideal modality to combine with a therapeutic HIV vaccine to reduce the number of latently infected CD4+ T cells in treated HIV-1 infected individuals.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection documented by previous HIV-1 serology or rapid test, or documented plasma HIV-1 RNA of >2000 copies/ml
* On stable cART regimen in accordance with the DHHS "Guidelines for the Use of Antiretroviral Agents in HIV-1-Infected Adults and Adolescents" with documented virologic suppression (VL<50 copies/ml) for ≥ 48 weeks.
* Baseline cell associated HIV-1 RNA is detectable (≥10copies/µg RNA)
* Laboratory values obtained within 30 days prior to study entry.

  * VL < 50 copies/ml
  * CD4+ T cell count > 500 cells/mm3
  * Absolute neutrophil count (ANC) ≥500/mm3
  * Hemoglobin ≥9.0 g/dL if female; 10 g/dL if male
  * Platelet count ≥75,000/mm3
  * AST (SGOT), ALT (SGPT) ≤3.5 × ULN
  * Alkaline phosphatase< 2.5 ULN
  * Total bilirubin ≤2.5 x ULN
  * Lipase ≤2.5 x ULN
  * Calculated creatinine clearance ≥70 mL/min as estimated by the Cockcroft-Gault equation:
* For men(140-age in yrs)x(body wt in kg)÷(serum creatinine in mg/dLx72)=CrCl (mL/min)*

  *For women, multiply the result by 0.85 = CrCl (mL/min)
* NOTE: A program to assist in calculations is available on the DMC web site at: http://www.fstrf.org/ACTG/ccc.html
* For women of reproductive potential, negative serum or urine pregnancy test
* Female candidates of reproductive potential is defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months) or have not undergone surgical sterilization (e.g., hysterectomy, or bilateral oophorectomy, or bilateral tubal ligation).
* Contraception requirements
* Female candidates of reproductive potential, who are participating in sexual activity that could lead to pregnancy, must agree that they will use at least two reliable barrier methods of contraception while receiving the protocol-specified treatments and for at least 24 weeks after completing stage I of the study.
* Men and women aged 18-55 years.
* Ability and willingness of subject to give written informed consent.
* Adequate venous access for phlebotomy

Exclusion Criteria:

* Previous immune based therapy
* History of vascular disease including h/o coronary artery disease, angina/MI, TIA/CVA, peripheral vascular disease/claudication
* Strong family history of cardiovascular disease
* Hyperlipidemia requiring medication
* Diabetes
* History of Tobacco use (≥10 pack years)
* HIV-related nephropathy
* History of vascular disease including history of coronary artery disease, angina/MI, TIA/CVA, peripheral vascular disease/claudication, poorly controlled hypertension
* Pregnancy or currently breast-feeding
* Desire to become pregnant during the course of study
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry.
* Known allergy/sensitivity to study drugs or their formulations.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* History of autoimmunity
* Chronic Hepatitis B (HepBSAg+) or C (HCV RNA positive)
* Current imprisonment or involuntary incarceration in a medical facility for psychiatric or physical (e.g., infectious disease) illness.
* Participation in any other clinical trial within 30 days prior to screening.
* Receipt of routine vaccination(s) within 7 days of study entry, or anticipated receipt of routine vaccination(s) during the first 4 weeks of the study. If routine vaccinations are to be administered following the first 4 weeks of the study, they cannot be administered within 7 days prior to weeks 16 and 48 follow up visits.
* Multi-drug resistant (MDR) HIV-1 precluding standard 3-drug therapy
* Any other clinical conditions or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07-26 (Actual); Study Completion 2016-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Study Director — Icahn School of Medicine at Mt. Sinai; Elizabeth Miller, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Martin Markowitz, MD, Principal Investigator — Aaron Diamond AIDS Research Center
Locations (1):
- The Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- [Background] Archin NM, Liberty AL, Kashuba AD, Choudhary SK, Kuruc JD, Crooks AM, Parker DC, Anderson EM, Kearney MF, Strain MC, Richman DD, Hudgens MG, Bosch RJ, Coffin JM, Eron JJ, Hazuda DJ, Margolis DM. Administration of vorinostat disrupts HIV-1 latency in patients on antiretroviral therapy. Nature. 2012 Jul 25;487(7408):482-5. doi: 10.1038/nature11286. PMID 22837004
- [Background] Shan L, Deng K, Shroff NS, Durand CM, Rabi SA, Yang HC, Zhang H, Margolick JB, Blankson JN, Siliciano RF. Stimulation of HIV-1-specific cytolytic T lymphocytes facilitates elimination of latent viral reservoir after virus reactivation. Immunity. 2012 Mar 23;36(3):491-501. doi: 10.1016/j.immuni.2012.01.014. Epub 2012 Mar 8. PMID 22406268
- [Background] Xing S, Bullen CK, Shroff NS, Shan L, Yang HC, Manucci JL, Bhat S, Zhang H, Margolick JB, Quinn TC, Margolis DM, Siliciano JD, Siliciano RF. Disulfiram reactivates latent HIV-1 in a Bcl-2-transduced primary CD4+ T cell model without inducing global T cell activation. J Virol. 2011 Jun;85(12):6060-4. doi: 10.1128/JVI.02033-10. Epub 2011 Apr 6. PMID 21471244
- [Background] Xing S, Siliciano RF. Targeting HIV latency: pharmacologic strategies toward eradication. Drug Discov Today. 2013 Jun;18(11-12):541-51. doi: 10.1016/j.drudis.2012.12.008. Epub 2012 Dec 25. PMID 23270785
- [Background] Elliot, J., et al. The Safety and Effect of Multiple Doses of Vorinostat on HIV Transcription in HIV+ Patients Receiving cART. in Conference on Retroviruses and Opportunistic Infections (CROI) (2013).
- [Background] Almeida M, Cordero M, Almeida J, Orfao A. Different subsets of peripheral blood dendritic cells show distinct phenotypic and functional abnormalities in HIV-1 infection. AIDS. 2005 Feb 18;19(3):261-71. PMID 15718836
- [Background] Almeida M, Cordero M, Almeida J, Orfao A. Persistent abnormalities in peripheral blood dendritic cells and monocytes from HIV-1-positive patients after 1 year of antiretroviral therapy. J Acquir Immune Defic Syndr. 2006 Apr 1;41(4):405-15. doi: 10.1097/01.qai.0000209896.82255.d3. PMID 16652047
- [Background] Almeida M, Cordero M, Almeida J, Orfao A. Abnormal cytokine production by circulating monocytes and dendritic cells of myeloid origin in ART-treated HIV-1+ patients relates to CD4+ T-cell recovery and HCV co-infection. Curr HIV Res. 2007 May;5(3):325-36. doi: 10.2174/157016207780636524. PMID 17504174
- [Background] Anthony DD, Yonkers NL, Post AB, Asaad R, Heinzel FP, Lederman MM, Lehmann PV, Valdez H. Selective impairments in dendritic cell-associated function distinguish hepatitis C virus and HIV infection. J Immunol. 2004 Apr 15;172(8):4907-16. doi: 10.4049/jimmunol.172.8.4907. PMID 15067070
- [Background] Buisson S, Benlahrech A, Gazzard B, Gotch F, Kelleher P, Patterson S. Monocyte-derived dendritic cells from HIV type 1-infected individuals show reduced ability to stimulate T cells and have altered production of interleukin (IL)-12 and IL-10. J Infect Dis. 2009 Jun 15;199(12):1862-71. doi: 10.1086/599122. PMID 19419334
- [Background] Chang JJ, Lacas A, Lindsay RJ, Doyle EH, Axten KL, Pereyra F, Rosenberg ES, Walker BD, Allen TM, Altfeld M. Differential regulation of toll-like receptor pathways in acute and chronic HIV-1 infection. AIDS. 2012 Mar 13;26(5):533-41. doi: 10.1097/QAD.0b013e32834f3167. PMID 22210629
- [Background] Fan Z, Huang XL, Kalinski P, Young S, Rinaldo CR Jr. Dendritic cell function during chronic hepatitis C virus and human immunodeficiency virus type 1 infection. Clin Vaccine Immunol. 2007 Sep;14(9):1127-37. doi: 10.1128/CVI.00141-07. Epub 2007 Jul 18. PMID 17634507
- [Background] Granelli-Piperno A, Golebiowska A, Trumpfheller C, Siegal FP, Steinman RM. HIV-1-infected monocyte-derived dendritic cells do not undergo maturation but can elicit IL-10 production and T cell regulation. Proc Natl Acad Sci U S A. 2004 May 18;101(20):7669-74. doi: 10.1073/pnas.0402431101. Epub 2004 May 5. PMID 15128934
- [Background] Hodges A, Sharrocks K, Edelmann M, Baban D, Moris A, Schwartz O, Drakesmith H, Davies K, Kessler B, McMichael A, Simmons A. Activation of the lectin DC-SIGN induces an immature dendritic cell phenotype triggering Rho-GTPase activity required for HIV-1 replication. Nat Immunol. 2007 Jun;8(6):569-77. doi: 10.1038/ni1470. Epub 2007 May 13. PMID 17496896
- [Background] Lester RT, Yao XD, Ball TB, McKinnon LR, Kaul R, Wachihi C, Jaoko W, Plummer FA, Rosenthal KL. Toll-like receptor expression and responsiveness are increased in viraemic HIV-1 infection. AIDS. 2008 Mar 30;22(6):685-94. doi: 10.1097/QAD.0b013e3282f4de35. PMID 18356597
- [Background] Majumder B, Janket ML, Schafer EA, Schaubert K, Huang XL, Kan-Mitchell J, Rinaldo CR Jr, Ayyavoo V. Human immunodeficiency virus type 1 Vpr impairs dendritic cell maturation and T-cell activation: implications for viral immune escape. J Virol. 2005 Jul;79(13):7990-8003. doi: 10.1128/JVI.79.13.7990-8003.2005. PMID 15956545
- [Background] Sabado RL, O'Brien M, Subedi A, Qin L, Hu N, Taylor E, Dibben O, Stacey A, Fellay J, Shianna KV, Siegal F, Shodell M, Shah K, Larsson M, Lifson J, Nadas A, Marmor M, Hutt R, Margolis D, Garmon D, Markowitz M, Valentine F, Borrow P, Bhardwaj N. Evidence of dysregulation of dendritic cells in primary HIV infection. Blood. 2010 Nov 11;116(19):3839-52. doi: 10.1182/blood-2010-03-273763. Epub 2010 Aug 6. PMID 20693428
- [Background] Shan M, Klasse PJ, Banerjee K, Dey AK, Iyer SP, Dionisio R, Charles D, Campbell-Gardener L, Olson WC, Sanders RW, Moore JP. HIV-1 gp120 mannoses induce immunosuppressive responses from dendritic cells. PLoS Pathog. 2007 Nov;3(11):e169. doi: 10.1371/journal.ppat.0030169. PMID 17983270
- [Background] Smed-Sorensen A, Lore K, Walther-Jallow L, Andersson J, Spetz AL. HIV-1-infected dendritic cells up-regulate cell surface markers but fail to produce IL-12 p70 in response to CD40 ligand stimulation. Blood. 2004 Nov 1;104(9):2810-7. doi: 10.1182/blood-2003-07-2314. Epub 2004 Jul 1. PMID 15231570
- [Background] Tan DB, Yong YK, Lim A, Tan HY, Kamarulzaman A, French M, Price P. Robust interferon-alpha and IL-12 responses by dendritic cells are related to efficient CD4+ T-cell recovery in HIV patients on ART. Clin Immunol. 2011 May;139(2):115-21. doi: 10.1016/j.clim.2011.02.015. Epub 2011 Feb 23. PMID 21429806
- [Background] Yonkers NL, Rodriguez B, Asaad R, Lederman MM, Anthony DD. Systemic immune activation in HIV infection is associated with decreased MDC responsiveness to TLR ligand and inability to activate naive CD4 T-cells. PLoS One. 2011;6(9):e23884. doi: 10.1371/journal.pone.0023884. Epub 2011 Sep 1. PMID 21912648
- [Background] Frleta D, Ochoa CE, Kramer HB, Khan SA, Stacey AR, Borrow P, Kessler BM, Haynes BF, Bhardwaj N. HIV-1 infection-induced apoptotic microparticles inhibit human DCs via CD44. J Clin Invest. 2012 Dec;122(12):4685-97. doi: 10.1172/JCI64439. Epub 2012 Nov 19. PMID 23160198
- [Background] Dillon SM, Robertson KB, Pan SC, Mawhinney S, Meditz AL, Folkvord JM, Connick E, McCarter MD, Wilson CC. Plasmacytoid and myeloid dendritic cells with a partial activation phenotype accumulate in lymphoid tissue during asymptomatic chronic HIV-1 infection. J Acquir Immune Defic Syndr. 2008 May 1;48(1):1-12. doi: 10.1097/QAI.0b013e3181664b60. PMID 18300699
- [Background] Butera ST, Roberts BD, Folks TM. Regulation of HIV-1 expression by cytokine networks in a CD4+ model of chronic infection. J Immunol. 1993 Jan 15;150(2):625-34. PMID 8380428
- [Background] Hoshino S, Konishi M, Mori M, Shimura M, Nishitani C, Kuroki Y, Koyanagi Y, Kano S, Itabe H, Ishizaka Y. HIV-1 Vpr induces TLR4/MyD88-mediated IL-6 production and reactivates viral production from latency. J Leukoc Biol. 2010 Jun;87(6):1133-43. doi: 10.1189/jlb.0809547. Epub 2010 Feb 9. PMID 20145198
- [Background] McNamara LA, Ganesh JA, Collins KL. Latent HIV-1 infection occurs in multiple subsets of hematopoietic progenitor cells and is reversed by NF-kappaB activation. J Virol. 2012 Sep;86(17):9337-50. doi: 10.1128/JVI.00895-12. Epub 2012 Jun 20. PMID 22718820
- [Background] Nabel G, Baltimore D. An inducible transcription factor activates expression of human immunodeficiency virus in T cells. Nature. 1987 Apr 16-22;326(6114):711-3. doi: 10.1038/326711a0. PMID 3031512
- [Background] Poli G, Kinter A, Justement JS, Kehrl JH, Bressler P, Stanley S, Fauci AS. Tumor necrosis factor alpha functions in an autocrine manner in the induction of human immunodeficiency virus expression. Proc Natl Acad Sci U S A. 1990 Jan;87(2):782-5. doi: 10.1073/pnas.87.2.782. PMID 2300561
- [Background] Saleh S, Wightman F, Ramanayake S, Alexander M, Kumar N, Khoury G, Pereira C, Purcell D, Cameron PU, Lewin SR. Expression and reactivation of HIV in a chemokine induced model of HIV latency in primary resting CD4+ T cells. Retrovirology. 2011 Oct 12;8:80. doi: 10.1186/1742-4690-8-80. PMID 21992606
- [Background] Tiemessen CT, Kilroe B, Martin DJ. Interleukin-8 fails to induce human immunodeficiency virus-1 expression in chronically infected promonocytic U1 cells but differentially modulates induction by proinflammatory cytokines. Immunology. 2000 Sep;101(1):140-6. doi: 10.1046/j.1365-2567.2000.00100.x. PMID 11012765
- [Background] Winckelmann, A., et al. Toll-like Receptor 9 Agonist Treatment Decreases the Proviral Reservoir in Peripheral Blood and Could Impact HIV-specific Immunity in Patients on cART. Conference on Retroviruses and Opportunistic Infections (CROI) (2013).
- [Background] Saleh S, Solomon A, Wightman F, Xhilaga M, Cameron PU, Lewin SR. CCR7 ligands CCL19 and CCL21 increase permissiveness of resting memory CD4+ T cells to HIV-1 infection: a novel model of HIV-1 latency. Blood. 2007 Dec 15;110(13):4161-4. doi: 10.1182/blood-2007-06-097907. Epub 2007 Sep 19. PMID 17881634
- [Background] Schulz O, Diebold SS, Chen M, Naslund TI, Nolte MA, Alexopoulou L, Azuma YT, Flavell RA, Liljestrom P, Reis e Sousa C. Toll-like receptor 3 promotes cross-priming to virus-infected cells. Nature. 2005 Feb 24;433(7028):887-92. doi: 10.1038/nature03326. Epub 2005 Feb 13. PMID 15711573
- [Background] Wille-Reece U, Flynn BJ, Lore K, Koup RA, Miles AP, Saul A, Kedl RM, Mattapallil JJ, Weiss WR, Roederer M, Seder RA. Toll-like receptor agonists influence the magnitude and quality of memory T cell responses after prime-boost immunization in nonhuman primates. J Exp Med. 2006 May 15;203(5):1249-58. doi: 10.1084/jem.20052433. Epub 2006 Apr 24. PMID 16636134
- [Background] Zhang Z, Kim T, Bao M, Facchinetti V, Jung SY, Ghaffari AA, Qin J, Cheng G, Liu YJ. DDX1, DDX21, and DHX36 helicases form a complex with the adaptor molecule TRIF to sense dsRNA in dendritic cells. Immunity. 2011 Jun 24;34(6):866-78. doi: 10.1016/j.immuni.2011.03.027. PMID 21703541
- [Background] Zhang Z, Yuan B, Lu N, Facchinetti V, Liu YJ. DHX9 pairs with IPS-1 to sense double-stranded RNA in myeloid dendritic cells. J Immunol. 2011 Nov 1;187(9):4501-8. doi: 10.4049/jimmunol.1101307. Epub 2011 Sep 28. PMID 21957149
- [Background] Akazawa T, Ebihara T, Okuno M, Okuda Y, Shingai M, Tsujimura K, Takahashi T, Ikawa M, Okabe M, Inoue N, Okamoto-Tanaka M, Ishizaki H, Miyoshi J, Matsumoto M, Seya T. Antitumor NK activation induced by the Toll-like receptor 3-TICAM-1 (TRIF) pathway in myeloid dendritic cells. Proc Natl Acad Sci U S A. 2007 Jan 2;104(1):252-7. doi: 10.1073/pnas.0605978104. Epub 2006 Dec 26. PMID 17190817
- [Background] Bogunovic D, Manches O, Godefroy E, Yewdall A, Gallois A, Salazar AM, Marie I, Levy DE, Bhardwaj N. TLR4 engagement during TLR3-induced proinflammatory signaling in dendritic cells promotes IL-10-mediated suppression of antitumor immunity. Cancer Res. 2011 Aug 15;71(16):5467-76. doi: 10.1158/0008-5472.CAN-10-3988. Epub 2011 Jul 5. PMID 21730023
- [Background] Longhi MP, Trumpfheller C, Idoyaga J, Caskey M, Matos I, Kluger C, Salazar AM, Colonna M, Steinman RM. Dendritic cells require a systemic type I interferon response to mature and induce CD4+ Th1 immunity with poly IC as adjuvant. J Exp Med. 2009 Jul 6;206(7):1589-602. doi: 10.1084/jem.20090247. Epub 2009 Jun 29. PMID 19564349
- [Background] Stahl-Hennig C, Eisenblatter M, Jasny E, Rzehak T, Tenner-Racz K, Trumpfheller C, Salazar AM, Uberla K, Nieto K, Kleinschmidt J, Schulte R, Gissmann L, Muller M, Sacher A, Racz P, Steinman RM, Uguccioni M, Ignatius R. Synthetic double-stranded RNAs are adjuvants for the induction of T helper 1 and humoral immune responses to human papillomavirus in rhesus macaques. PLoS Pathog. 2009 Apr;5(4):e1000373. doi: 10.1371/journal.ppat.1000373. Epub 2009 Apr 10. PMID 19360120
- [Background] Tewari K, Flynn BJ, Boscardin SB, Kastenmueller K, Salazar AM, Anderson CA, Soundarapandian V, Ahumada A, Keler T, Hoffman SL, Nussenzweig MC, Steinman RM, Seder RA. Poly(I:C) is an effective adjuvant for antibody and multi-functional CD4+ T cell responses to Plasmodium falciparum circumsporozoite protein (CSP) and alphaDEC-CSP in non human primates. Vaccine. 2010 Oct 21;28(45):7256-66. doi: 10.1016/j.vaccine.2010.08.098. Epub 2010 Sep 21. PMID 20846528
- [Background] Vagenas P, Aravantinou M, Williams VG, Jasny E, Piatak M Jr, Lifson JD, Salazar AM, Blanchard JL, Gettie A, Robbiani M. A tonsillar PolyICLC/AT-2 SIV therapeutic vaccine maintains low viremia following antiretroviral therapy cessation. PLoS One. 2010 Sep 21;5(9):e12891. doi: 10.1371/journal.pone.0012891. PMID 20877632
- [Background] Zobywalski A, Javorovic M, Frankenberger B, Pohla H, Kremmer E, Bigalke I, Schendel DJ. Generation of clinical grade dendritic cells with capacity to produce biologically active IL-12p70. J Transl Med. 2007 Apr 12;5:18. doi: 10.1186/1479-5876-5-18. PMID 17430585
- [Background] Checkley Luttge, M., et al. Natural Killer Cells Can Target and Eliminate Latently HIV-1-Infected Primary T cells following Proviral Reactivation. Conference on Retroviruses and Opportunistic Infections (CROI) (2013).
- [Background] Caskey M, Lefebvre F, Filali-Mouhim A, Cameron MJ, Goulet JP, Haddad EK, Breton G, Trumpfheller C, Pollak S, Shimeliovich I, Duque-Alarcon A, Pan L, Nelkenbaum A, Salazar AM, Schlesinger SJ, Steinman RM, Sekaly RP. Synthetic double-stranded RNA induces innate immune responses similar to a live viral vaccine in humans. J Exp Med. 2011 Nov 21;208(12):2357-66. doi: 10.1084/jem.20111171. Epub 2011 Nov 7. PMID 22065672
- [Background] Okada H, Kalinski P, Ueda R, Hoji A, Kohanbash G, Donegan TE, Mintz AH, Engh JA, Bartlett DL, Brown CK, Zeh H, Holtzman MP, Reinhart TA, Whiteside TL, Butterfield LH, Hamilton RL, Potter DM, Pollack IF, Salazar AM, Lieberman FS. Induction of CD8+ T-cell responses against novel glioma-associated antigen peptides and clinical activity by vaccinations with alpha-type 1 polarized dendritic cells and polyinosinic-polycytidylic acid stabilized by lysine and carboxymethylcellulose in patients with recurrent malignant glioma. J Clin Oncol. 2011 Jan 20;29(3):330-6. doi: 10.1200/JCO.2010.30.7744. Epub 2010 Dec 13. PMID 21149657
- [Background] Poly-ICLC Investigational Brochure (Hiltonol®, Oncovir).
- [Background] Trumpfheller C, Longhi MP, Caskey M, Idoyaga J, Bozzacco L, Keler T, Schlesinger SJ, Steinman RM. Dendritic cell-targeted protein vaccines: a novel approach to induce T-cell immunity. J Intern Med. 2012 Feb;271(2):183-92. doi: 10.1111/j.1365-2796.2011.02496.x. Epub 2012 Jan 4. PMID 22126373
- [Background] Marcus PI, Sekellick MJ. Combined sequential treatment with interferon and dsRNA abrogates virus resistance to interferon action. J Interferon Cytokine Res. 2001 Jun;21(6):423-9. doi: 10.1089/107999001750277907. PMID 11440640
- [Derived] Saxena M, Sabado RL, La Mar M, Mohri H, Salazar AM, Dong H, Correa Da Rosa J, Markowitz M, Bhardwaj N, Miller E. Poly-ICLC, a TLR3 Agonist, Induces Transient Innate Immune Responses in Patients With Treated HIV-Infection: A Randomized Double-Blinded Placebo Controlled Trial. Front Immunol. 2019 Apr 9;10:725. doi: 10.3389/fimmu.2019.00725. eCollection 2019. PMID 31024557

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Poly-ICLC: Poly-ICLC: Poly-ICLC (Hiltonol®, Oncovir) Administration - On days 1 and 2, patients randomized to this arm will be injected subcutaneously in the arm with 1.4 mg of Poly-ICLC (Hiltonol®, Oncovir). Each subject will receive a total of 2 SC doses of Poly-ICLC. The volume of each injection is 0.7ml.
- Arm B: Normal Saline: Normal Saline: Normal Saline - On days 1 and 2, patients randomized to this arm will be injected subcutaneously in the arm with normal saline obtained from the Rockefeller University Pharmacy. Each subject will receive a total of 2 SC doses of normal saline. The volume of each injection is 0.7ml.
Period: Overall Study
Arm/Group | Arm A: Poly-ICLC | Arm B: Normal Saline
Started | 12 | 3
Completed | 12 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Poly-ICLC | Arm B: Normal Saline | Total
Number analyzed (Participants) | 12 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (9.32) | 34.33 (4.03) | 39.73 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number Participants With Adverse Events
Description: Safety measured by number of participants with adverse events.
Time Frame: Up to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Poly-ICLC | Arm B: Normal Saline
Number analyzed (Participants) | 12 | 3
Participants | 11 | 3

2. Secondary Outcome: Plasma Interferon-gamma-inducible Protein-10 (IP-10) Level
Description: One of the biomarkers of cellular immune activation and exhaustion quantified by flow cytometry. Normal range is 7.8-500 pg/ml.
Time Frame: Day 2 and Day 4
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Arm A: Poly-ICLC | Arm B: Normal Saline
Number analyzed (Participants) | 12 | 3
pg/ml
  Day 2 | 381.43 (187.67) | 100.65 (13.5)
  Day 4 | 450.51 (144.9) | 139.39 (42.74)

3. Secondary Outcome: CD8 CD38 (Mean of Fluorescence)
Description: the CD38-activation marker on CD8 T-cells (CD8/CD38).
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: mean fluorescent intensity (MFI)
Arm/Group | Arm A: Poly-ICLC | Arm B: Normal Saline
Number analyzed (Participants) | 12 | 3
mean fluorescent intensity (MFI) | 8.69 (6.77) | 2.35 (2.27)

4. Secondary Outcome: NK Cell Number
Description: Natural killer cells or NK cells are part of the innate immune defense against infection and cancer.
Time Frame: at 48 weeks
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Arm A: Poly-ICLC | Arm B: Normal Saline
Number analyzed (Participants) | 12 | 3
cells/µL | 20.68 (16.06) | 19.41 (15.45)

5. Secondary Outcome: Percent Change in CD4+ Tcell-associated HIV-1 RNA as Compared to Baseline
Description: CD4+ Tcell-associated HIV-1 RNA to determine whether Poly-ICLC disrupts viral latency in HIV-1-infected individuals on anti-retroviral therapy.Viral transcription assessed by monitoring cell associated HIV-1 RNA. Percent change compared to baseline.
Time Frame: Baseline, Day 2, Day 4, Day 8, Day 28
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm A: Poly-ICLC | Arm B: Normal Saline
Number analyzed (Participants) | 12 | 3
percent change
  Day 2 | 102.8 (30.65) | 186.3 (163.4)
  Day 4 | 134.8 (90.3) | 254.7 (223.8)
  Day 8 | 161.0 (112.3) | 66.33 (22.74)
  Day 28 | 199.6 (247.2) | 126.7 (65.77)

ADVERSE EVENTS:
Arm/Group | Arm A: Poly-ICLC | Arm B: Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/3
Serious Adverse Events (participants affected / at risk) | 11/12 | 3/3
Other Adverse Events (participants affected / at risk) | 1/12 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Poly-ICLC (N=12) | Arm B: Normal Saline (N=3)
Chills (General disorders) | 3 | 0
erythema (Surgical and medical procedures) | 5 | 0 — Injection site reaction
Pain (Surgical and medical procedures) | 10 | 0 — Injection site reaction
Fatigue (General disorders) | 7 | 3
Fever (General disorders) | 4 | 0
Malaise (General disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 2
Myalgias (Musculoskeletal and connective tissue disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Poly-ICLC (N=12) | Arm B: Normal Saline (N=3)
Low neutrophils count (Blood and lymphatic system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Small sample size, gender homogeneity, and exclusion of older individuals (>55 years) and common comorbidities such as cardiovascular disease and diabetes limit the generalizability of the safety findings in the HIV-infected population as a whole.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes